CLINICAL TRIAL: NCT01541189
Title: A 8-week, Multi Center(10),Single Arm, Open-labeled Prospective Study of Valsartan 160 mg in 200 Mild to Moderate Chinese Hypertension Patients Forced Titrated From 2-week Therapy of Valsartan 80 mg.
Brief Title: Double-dose Valsartan Monotherapy in Hypertension Treatment: an Effectiveness and Safety Evaluation in Chinese Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489ACN14
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
Keywords: hypertension; valsartan
MeSH Terms: conditions — Hypertension | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- valsartan (Experimental): After 1-week screening period, all of the eligible patients receive valsartan 80mg/day for 2 weeks, then the dosage will be titrated to 160mg/day for further 8 weeks therapy for all of the subjects.
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Valsartan — 80 mg/day for 2 weeks, up-titrated to 160 mg/day for further 8 weeks

SUMMARY:
To evaluate efficacy and safety of valsartan 160mg in Chinese hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Naive primary hypertension patients or primary hypertensive patients on mono antihypertensive therapy:
* All treatment-naive patients need to have 140mmHg≤MSSBP<180mmHg and 90mmHg≤MSDBP< 110mmHg at visit 1
* For patients on mono antihypertensive therapy, MSSBP/MSDBP should <160/100mmHg at visit 1 (the beginning of screening period); and at visit 2(the beginning of theraputic period), they should have MSSBP≥140 mmHg and <180mmHg AND MSDBP≥90 mmHg and <110mmHg

Exclusion Criteria:

* Severe hypertension
* Malignant hypertension
* Secondary hypertension
* Renal dysfunction(serum creatinine > 2.0mg(176.8μmol/L)at visit 1)
* Hepatic disease
* History of hypertensive encephalopathy or cerebrovascular accident within 6 months
* History of myocardial infarction, coronary revascularization within 6 months
* Type 1 diabetes mellitus
* patietns with HbA1c >8% at visit 1
* Women in pregnancy and lactation
* Potentially fertile female patients not using effective contraceptive methods
* Be allergy to study drug.

Other protocol defined inclusion/exlusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline and week 2 in blood pressure at week 10 | Baseline, 2 week and 10 weeks

SECONDARY OUTCOMES:
Percentage of of patients who achieve BP<140/90mmHg | Baseline and 10 weeks
Change from baseline in ABPM (Ambulatory Blood Pressure Monitor) at week 10 | Baseline and 10 weeks
  Each subject will receive 24-hour ABPM at baseline and week 10.
Change from baseline in HBPM (Home Blood Pressure Monitor) at week 10 | Baseline and 10 weeks
  Each subject will receive HBPM at baseline, week 2, week 6 and week 10 respectively.For baseline HBPM, it was performed in the evening before visit 2 and in the morning of visit 2(before intake of study drug). in terms of the following 3 times of HBPM, they are performed during 5 days before each visit.
Number of patients with adverse events, serious adverse events | during 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Beijing, Beijing Municipality, China